CLINICAL TRIAL: NCT02448095
Title: Ponatinib Survey: Retrospective Evaluation of CML Patients in the National Compassionate Program According to the 648/96 Decree
Brief Title: Retrospective Evaluation of CML Patients in the National Compassionate Program
Status: Terminated | Type: Observational
Why Stopped: lack of interest
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: CML1214
Record Dates: First submitted 2015-05-15; First posted 2015-05-19 (Estimated); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Chronic Myeloid Leukemia; Philadelphia Positive
Keywords: Chronic myeloid leukemia; Philadelphia positive; Compassionate use
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — ponatinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CML ph+ patients: Chronic myeloid leukemia patients who are philadelphia positive
  Interventions: Drug: Ponatinib

INTERVENTIONS:
Drug: Ponatinib — Observation of tolerability and safety profiles

SUMMARY:
This observational study aims at assessing the tolerability and safety profiles of Ponatinib, a drug used for Chronic Myeloid Leukemia patients who are Philadelphia positive. This drug is used during the chronic phase of the disease, according to the Italian national compassionate law 648/96.

DETAILED DESCRIPTION:
This observational study aims at assessing the tolerability and safety profiles of Ponatinib, a drug used for Chronic Myeloid Leukemia patients who are Philadelphia positive. This drug is used during the chronic phase of the disease, according to the Italian national compassionate law 648/96.

ELIGIBILITY:
Inclusion Criteria:

* CML Ph+ patients in chronic phase
* 18 years old or older
* Patients have received either Dasatinib or Nilotinib and resulted resistant or not tolerant to the drugs or have developed the T3151 mutation
* Patients have started Ponatinib at least 12 months before registration
* Informed consent signed at registration

Exclusion Criteria:

* CML Ph+ patients in accelerated or blast phase with acute lymphoblastic leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CML Ph+ patients in the Ponatinib compassionate use program
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | Maximum of 60 months from treatment start
  General adverse events and grade 3-4 adverse events according to NCI CTCAE version 4.0

SECONDARY OUTCOMES:
Number of patients with hematological complete response | Maximum of 60 months from treatment start
  Hematological complete response and related responses, such as major cytogenetic response, complete cytogenetic response and major molecular response.
Number of days from treatment start till response | Maximum of 60 months from treatment start
Total number of patients alive | 12 months after patient enrollment in the study
  Overall survival
Number of patients in event free survival | 12 months after patient enrollment in the study
  Event free survival
Number of patients in progression free survival | 12 months after patient enrollment in the study
  Progression free survival
Number of mutations | Maximum of 60 months from treatment start
  Both at the beginning and at the end of treatment
Number of units of Ponatinib administered per units of time | Maximum of 60 months from treatment start
  Chemotherapy dose intensity represents unit dose of chemotherapy administered per unit time.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Fava, Study Chair — Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2 - Orbassano
Locations (10):
- Italy (10):
  - UO Ematologia con trapianto-Università degli Studi di Bari Aldo Moro, Bari
  - IRCCS_AOU San Martino-IST.Clinica Ematologica, Genova
  - ASL Le/1 P.O. Vito Fazzi - U.O. di Ematologia ed UTIE, Lecce
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico UOC Oncoematologia- Padiglione Marcora 2° piano, Milan
  - Azienda Ospedaliera "S.Gerardo", Monza
  - S.C.D.U. Ematologia - DIMECS e Dipartimento Oncologico - Università del Piemonte Orientale Amedeo Avogadro, Novara
  - Dip. di Scienze Cliniche e Biologiche - Ospedale S. Luigi Gonzaga-Medicina Interna 2 - Orbassano, Orbassano
  - S.C. Ematologia - Fondazione IRCCS Policlinico S. Matteo, Pavia
  - Dipartimento Emato-Oncologia A.O."Bianchi-Melacrino-Morelli", Reggio Calabria
  - U.O.C. Ematologia - Ospedale S. Eugenio, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: GIMEMA Foundation website — http://www.gimema.it